CLINICAL TRIAL: NCT05210907
Title: A Phase Ib, Clinical Trial of Hospital-manufactured CD19 Chimeric Antigen Receptor T Cells (SNUH-CD19-CAR-T) in Children and Adolescents With Relapsed or Refractory CD19 Positive Acute Lymphoblastic Leukemia
Brief Title: Clinical Study of Hospital-manufactured CD19 CAR-T in Children and Adolescents With Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH_CART_CD19ALL
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR-T therapy (Experimental): SNUH-CD19-CAR-T is administered as an intravenous infusion.
  Interventions: Biological: SNUH-CD19-CAR-T

INTERVENTIONS:
Biological: SNUH-CD19-CAR-T — SNUH-CD19-CAR-T is an autologous CAR-T from T cells collected from each patient. Administer a single dose of SNUH-CD19-CAR-T to patients with relapsed or refractory CD19 positive B-cell acute lymphoblastic leukemia, and evaluate safety and efficacy of SNUH-CD19-CAR-T for 12 months after the infusion.

SUMMARY:
Chimeric antigen receptor T cells (CAR-T cells) have been developed to treat relapsed and refractory hematological malignancies with promising outcome in patients with very poor prognosis. The purpose of this clinical study is to produce the CD19[cluster of differentiation antigen 19] CAR-T (SNUH-CD19-CAR-T) at the investigational site and to evaluate safety and efficacy of SNUH-CD19-CAR-T in children and adolescent with relapsed/refractory B-cell acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Relapsed or refractory CD19 Positive Acute Lymphoblastic Leukemia. All subjects must be younger than 26 years old at the time of obtaining informed consent

  a. 2nd or greater BM[bone marrow] relapse OR b. Any BM relapse after allogeneic SCT[stem cell transplant] and must be ≥ 6 months from SCT at the time of SNUH_CD19_CAR-T infusion OR c .Refractory as defined by not achieving a CR after 2 cycles of a standard chemotherapy regimen or chemorefractory as defined by not achieving a CR after 1 cycle of standard chemotherapy for relapsed leukemia OR d. Ineligible for allogeneic SCT because of:
  * Severe comorbid disease
  * Other contraindications to allogeneic SCT conditioning regimen
  * Lack of suitable donor

    2. Documentation of CD19 tumor expression in bone marrow or peripheral blood by flow cytometry.

    3. Karnofsky (age ≥ 16 years) or Lansky (age < 16 years) performance status ≥ 50 at screening

Exclusion Criteria:

1. Evidence of uncontrolled hepatitis B virus (HBV) or hepatitis C virus (HCV) based on assessment done by treating physicians.
2. Known human immunodeficiency virus (HIV) infection.
3. Presence of clinically active uncontrolled infection based on assessment done by treating physicians. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of progression are present. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
4. Pregnant or nursing (lactating) women.

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and its severity | 12 months post SNUH-CD19-CAR-T infusion

SECONDARY OUTCOMES:
Patients with CR[complete remission] after Hospital-manufactured CAR-T infusion | 1 month post SNUH-CD19-CAR-T infusion
Overall survival and event-free survival | 12 months post SNUH-CD19-CAR-T infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided